CLINICAL TRIAL: NCT01635920
Title: A Comparison of Silicone Hydrogel Lenses: Colored Versus Non-Colored
Brief Title: A Comparison of Silicone Hydrogel Contact Lenses: AIR OPTIX® COLORS Versus AIR OPTIX® AQUA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: C-12-004
Record Dates: First submitted 2012-07-05; First posted 2012-07-10 (Estimated); Results first posted 2014-03-28 (Estimated); Last update posted 2014-03-28 (Estimated); Status verified 2014-02

CONDITIONS: Myopia
Keywords: contact lenses; color contact lenses; myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- AIR OPTIX® COLORS (Experimental): Lotrafilcon B contact lens with color worn bilaterally for a minimum of 5 days per week, 8 hours per day, in daily wear modality for 4 weeks.
  Interventions: Device: Lotrafilcon B contact lens with color
- AIR OPTIX® AQUA (Active Comparator): Lotrafilcon B contact lens worn bilaterally for a minimum of 5 days per week, 8 hours per day, in daily wear modality for 4 weeks.
  Interventions: Device: Lotrafilcon B contact lens

INTERVENTIONS:
Device: Lotrafilcon B contact lens with color — Silicone hydrogel contact lens with color
  Other Names: AIR OPTIX® COLORS
  Arms: AIR OPTIX® COLORS
Device: Lotrafilcon B contact lens — Silicone hydrogel contact lens
  Other Names: AIR OPTIX® AQUA
  Arms: AIR OPTIX® AQUA

SUMMARY:
The purpose of this study was to compare the overall fit of AIR OPTIX® COLORS to AIR OPTIX® AQUA contact lenses.

DETAILED DESCRIPTION:
Eligible participants were randomized at Visit 1 (Screening) to receive 1 of the 2 investigational products (1:1 assignment). Between Visit 1 and Visit 2, participants wore their habitual AIR OPTIX® AQUA lenses. Investigational products were dispensed at Visit 2 (Baseline), after which participants were asked to return for 2 additional visits: Visit 3 (Day 14) and Visit 4 (Day 28).

ELIGIBILITY:
Inclusion Criteria:

* Visual acuity of at least 20/30 (Snellen) in each eye at distance with contact lenses and best corrected visual acuity ≥ 20/25 in each eye.
* Manifest cylinder less than or equal to 0.75 diopter (D) (within the previous year) in each eye.
* Successful wear of AIR OPTIX® AQUA soft contact lenses in both eyes during the past 3 months for a minimum of 5 days per week and 8 hours per day.
* Willing to sign an Informed Consent form. If under legal age of consent, legally authorized representative must also sign an Informed Consent form.
* Other protocol-specified inclusion criteria may apply.

Exclusion Criteria:

* Any ocular or systemic medical condition that may, in the opinion of the investigator, preclude safe administration of the test articles or affect the results of this study.
* Wears habitual lenses in an extended wear modality (sleeping in lenses overnight / not removing lenses on a daily basis).
* Monovision, monocular (only one eye with functional vision), or fit with only one lens.
* History of intolerance or hypersensitivity to any component of the test articles.
* Use of any over-the-counter (OTC) or prescribed topical ocular medications within previous 7 days (excluding rewetting drops).
* Moderate or severe corneal edema, corneal vascularization, corneal staining, injection, tarsal abnormalities, "other" complications, and any corneal infiltrates.
* Current or history of ocular infection, severe inflammation, or disease within previous 6 months.
* Any systemic disease that may affect the eye or be exacerbated by use of contact lenses or contact lens solutions.
* Ocular or intra-ocular surgery within the previous 12 months (excluding placement of punctal plugs).
* Use of medications contributing to dry eye or ocular irritation unless on a stable dosing regimen for a minimum of 30 days prior to study entry and able to remain on stable regimen throughout the study.
* Participation in any investigational clinical study within previous 30 days.
* Other protocol-specified exclusion criteria may apply.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 258 (Actual)
Dates: Start 2012-06; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Holden Thomas, O.D., Study Director — Alcon Research

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 15 study centers located in the United States.
Pre-assignment Details: Of the 258 participants enrolled, 7 participants did not receive study lenses. This reporting group includes all enrolled and randomized participants who received study lenses (251).
Period: Overall Study
Arm/Group | AIR OPTIX® COLORS | AIR OPTIX® AQUA
Started | 125 | 126
Completed | 122 | 125
Not Completed | 3 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Subject decision | 2 | 0

BASELINE CHARACTERISTICS:
Population: The analysis population includes all enrolled and randomized participants who received study lenses (251).
Groups:
- Total: Total of all reporting groups
Arm/Group | AIR OPTIX® COLORS | AIR OPTIX® AQUA | Total
Number analyzed (Participants) | 125 | 126 | 251
Age, Customized [Number; unit: participants]
  16-17 years | 10 | 5 | 15
  18-64 years | 115 | 119 | 234
  ≥ 65 years | 0 | 2 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 92 | 91 | 183
  Male | 33 | 35 | 68

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Same Fit in Both Eyes
Description: Lens fit was assessed by the investigator for each eye using a biomicroscope (slit lamp), which magnifies the appearance of the contact lens on the participant's eye. Lens fit was graded on a 5-point scale, with 2=unacceptably loose, 1=acceptably loose, 0=optimal, -1=acceptably tight, and -2=unacceptably tight. "Same fit" was defined as an eye that achieved an acceptable or optimal overall lens fit with the study lens, that was also within one grade of the value observed on the same eye with the habitual lens at the baseline visit.
Time Frame: Up to Day 28
Population: ITT: All enrolled and dispensed participants who had at least one study visit after being dispensed with study lenses (N=125,126). No imputation was used for the missing values. Here, "n" is the number of participants with non-missing values at the specific time point for each arm group, respectively.
Measure: Number; unit: percentage of participants
Arm/Group | AIR OPTIX® COLORS | AIR OPTIX® AQUA
Number analyzed (Participants) | 125 | 126
percentage of participants
  Day 14 (n=121,126) | 99.2 | 100
  Day 28 (n=122, 124) | 99.2 | 99.2

2. Secondary Outcome: Subjective Rating of Overall Comfort
Description: Overall comfort, as rated by the participant on a 10-point scale, with 1 being poor and 10 being excellent. The participant rated both eyes together by providing one single rating.
Time Frame: Up to Day 28
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- AIR OPTIX® COLORS: Lotrafilcon B contact lens with print worn bilaterally for a minimum of 5 days per week, 8 hours per day, in daily wear modality for 4 weeks.
Arm/Group | AIR OPTIX® COLORS | AIR OPTIX® AQUA
Number analyzed (Participants) | 125 | 126
units on a scale
  Day 14 (n=122, 126) | 8.4 (1.8) | 8.9 (1.3)
  Day 28 (n=122, 125) | 8.5 (1.4) | 8.9 (1.4)

ADVERSE EVENTS:
Time Frame: Adverse Events (AE) were collected after signing the informed consent, and reported for the duration of the study (2 months).
Description: AEs were defined as any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users or other persons, whether or not related to the investigational medical device. The analysis population includes all enrolled and randomized participants who received study lenses.
Arm/Group | AIR OPTIX® COLORS | AIR OPTIX® AQUA
Serious Adverse Events (participants affected / at risk) | 0/125 | 0/126
Other Adverse Events (participants affected / at risk) | 0/125 | 0/126

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.